CLINICAL TRIAL: NCT00820430
Title: A Multi-Center Trial on MR Image Markers of Knee Articular Cartilage Damage in Osteoarthritis
Brief Title: MRI Markers of Cartilage Damage in Knee With Osteoarthritis
Status: Completed | Type: Observational
Sponsor: American College of Radiology (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: ACRIN PA 4001; SAP #4100026182
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee
Keywords: osteoarthritis; knee; magnetic resonance imaging; knee cartilage; reproducibility
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Control--Non-Osteoporotic Knee: Kellgren-Lawrence (KL) scale score of 0, Age: 18-35 years
  Interventions: Other: Magnetic Resonance Imaging
- Minimal Osteoarthritis, Knee: Kellgren-Lawrence (KL) scale score of 1 or 2, Age: Older than 18; no upper limit
  Interventions: Other: Magnetic Resonance Imaging
- Moderate Osteoarthritis, Knee: Kellgren-Lawrence (KL) scale score of 3, Age: Older than 18; no upper limit
  Interventions: Other: Magnetic Resonance Imaging

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Subjects will undergo 4 sequential MRI evaluations of the target knee within a 4 week period to calculate precision error (ICC) in determination of cartilage morphometry (cartilage volume, mean thickness, and surface area), cartilage collagen (regional cartilage T2), and cartilage proteoglycan (regional cartilage T1rho).
  Other Names: MRI; knee MRI; knee magnetic resonance imaging

SUMMARY:
The objectives of this study are: to identify and develop techniques to minimize precision errors in magnetic resonance imaging (MRI) evaluation of knee cartilage, and to determine if results from newly-identified MRI techniques in measuring cartilage changes and structure can be reproduced.

DETAILED DESCRIPTION:
The development of a disease modifying osteoarthritis drugs (DMOADs) is currently limited by the inability to detect and monitor early cartilage damage that would be amenable to treatment. There is growing interest within the pharmaceutical and research community to use Magnetic Resonance Imaging (MRI) to identify biochemical and structural changes in the cartilage extra cellular matrix that occur early in the disease process. Although these techniques have been validated in small studies at single sites, multi-center evaluation of accuracy and precision, needed to apply these techniques to clinical trials of DMOADs, has not been performed. To address this need, the primary objective for this protocol is to identify and develop techniques to minimize systematic errors that decrease precision of MRI evaluation of knee cartilage, and to assess the reproducibility of the newly identified MRI techniques in measuring the cartilage morphometry and structure. Successful completion of this project may establish a multi-center imaging network in Pennsylvania for MRI evaluation of potential disease modifying osteoarthritis drugs (DMOADs) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >18 years old;
* Participants must have a KL score between 0 and 3;
* Participants must have clearance to use protocol specified equipment: 3T MRI with parallel imaging capability and phased array knee coil (minimum 4 elements);
* Participant had no change of treatment occur within the last 6 months;
* Participants have no plans of changing to a different treatment within the next 3 months;
* Participant must provide a study-specific signed informed consent form.

Exclusion Criteria:

* Patients with contraindication to 3T MRI: Claustrophobia, Implanted metal or medical device that is not approved for MRI scanning at 3T, pregnancy, inability to tolerate relative immobility for 1 hour;
* Patients with prior knee surgery or trauma of the knee;
* Patients with KL score of 4.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This multi-center trial comprises only facilities within Pennsylvania. Study participants for the normal cohorts will be recruited through print flyers. It is anticipated that the study participants with mild to moderate OA will be identified by the radiologists interpreting the knee x-rays.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary study goals are to develop and evaluate MRI techniques that minimize systematic errors in measuring knee cartilage, and to assess the reproducibility of MRI techniques comparing normal and osteoarthritic knees across institutions. | 4 sequental MRI evaluations of the target knee within a 4-week period

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Mosher, MD, Principal Investigator — Milton S. Hershey Medical Center; Ravinder Reddy, PhD, Study Chair — University of Pennsylvania, MMRRCC
Locations (5):
- United States (5):
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania